CLINICAL TRIAL: NCT00701909
Title: The Effectiveness of Small Doses of Ketamine With Morphine on Decreasing Pain Responses During Open Wound Care
Brief Title: Pain Medicine for Wound Care Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H2280-32187-01
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Wound Care; Pain Intensity; Hyperalgesia; Nausea; Vomiting; Hallucinations
Keywords: wound care; procedural pain intensity; procedural hyperalgesia; wound care pain intensity; wound care hyperalgesia; Wound care pain quality; Level of drowsiness; level of nausea; Level of vomiting; Level of hallucinations; Level of dysphoria
MeSH Terms: conditions — Pain; Hyperalgesia; Nausea; Vomiting; Hallucinations | interventions — Morphine; Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine plus Ketamine, then Morphine plus Saline (placebo) (Active Comparator): During the first wound care procedure, patients received morphine 0.05 mg/kg (a maximum dose of 4 mg) plus ketamine 0.25 mg/kg (MK). Then, during the second wound care procedure, patients received morphine 0.1 mg/kg (a maximum dose of 8 mg) plus saline (MS).
  Interventions: Drug: Morphine plus Ketamine; Drug: Morphine plus Saline (placebo)
- Morphine plus Saline (placebo), then Morphine plus Ketamine (Placebo Comparator): During the first wound care procedure, patients received morphine 0.1 mg/kg (a maximum dose of 8 mg) plus saline (MS). Then, during the second wound care procedure, patients received morphine 0.05 mg/kg (a maximum dose of 4mg) plus ketamine 0.25 mg/kg (MK)
  Interventions: Drug: Morphine plus Ketamine; Drug: Morphine plus Saline (placebo)

INTERVENTIONS:
Drug: Morphine plus Ketamine — Morphine 0.05 mg/kg (maximum dose of 4 mg) IV plus Ketamine 0.25 mg/kg IV. Then, Morphine 0.1 mg/kg (maximum dose of 8 mg) IV plus Saline IV
Drug: Morphine plus Saline (placebo) — Morphine 0.1 mg/kg (maximum dose of 8 mg) IV plus Saline IV. Then, Morphine 0.05 mg/kg (maximum dose of 4 mg) IV plus Ketamine 0.25 mg/kg IV.

SUMMARY:
This is a randomized double-blind study to determine if the administration of a small-dose of ketamine (an anesthetic)added to morphine (an opioid) contributes to reducing pain intensity during open wound care procedure (WCP)in patients who have had a traumatic injury and are in an Intensive Care Unit. Patients will be randomized to receive morphine plus saline (a placebo) or morphine plus ketamine before the WCP. The second time the patient is scheduled for WCP (no less than 24 hours), patients will be crossed over to receive the treatment they did not receive the first time. It is hypothesized that patients who receive the combination of morphine and ketamine will have better pain control during the procedure than patients who just receive morphine.

DETAILED DESCRIPTION:
An open wound care procedure causes pain and sometimes the use of medication such as morphine alone does not adequately help to alleviate pain during this procedure. This study is being done to learn if the administration of another medication named ketamine by the vein in addition to morphine is more effective in alleviating pain during the wound cleansing procedure than the administration of morphine alone. Patients will be eligible for the study if they are 21 years and older, have an open surgical or traumatic wound with a duration of no more than 10 days, had a wound pain intensity score more than 3 in a scale of 0 to 10 where 0 is no pain and 10 is the worst pain imaginable during a previous wound care procedure, and have an intravenous access.

A total of 50 patients with these same characteristics are expected to take part in this study. Patients who agree to take part in this study will, one day, receive receive an injection via the vein of morphine 0.05 mg per kilogram of their weight (maximum dose of 4 mg) and another of ketamine 0.25 mg per kilogram of their weight prior receiving the wound care procedure and, on the other day, will receive an injection via the vein of morphine 0.1 mg per kilogram of their weight (maximum dose of 8 mg) and another of saline prior receiving the wound care procedure. They will not be able to know if they receive ketamine or saline the first time or second time.

Ketamine is a drug approved by the U.S. Food and Drug Administration (FDA) for anesthesia but not approved to provide analgesia (relieve pain). However, small doses of ketamine are used (out of its indications) in the clinical area to provide analgesia, and its analgesic properties have been studied by many researchers.

Before the wound care procedure subjects will be asked to rate their wound pain intensity at rest at that moment and in the past 24 hours (including "worst" and "average" pain), overall pain intensity at rest at this moment and "worst" and "average" in the past 24 hours using a 0 to 10 scale where 0 is no pain and 10 is the worst pain imaginable. They will be given a list of common words that might describe their pain, and a body outline to indicate where the pain is. In addition, they will be asked to rate their level of sleepiness using a 0 to 10 scale where 0 is not at all sleepy and 10 is extremely sleepy.

After removing the outer dressing, patients will be tested for pain sensitivity around the wound with a thin, short length of plastic (like a little straw), which will be pressed against their skin from the outside of the wound towards the wound and they will be asked to report a distinct change in perception. The first point where a "painful", "sore", or "sharper" feeling occurs will be marked in the skin to measure the distance of this mark to the wound. If no change in perception occurs, stimulation will be stopped 0.5 cm from the wound. This measure is experimental.

Immediately after the wound care procedure the following will be measured: (1) "worst" wound pain intensity experienced during the wound care procedure, (2) description of pain quality during the wound care procedure, (3) level of sleepiness, (4) side effects such as unpleasant sensation will be measured using a 0 to 10 scale, where 0 means no unpleasant sensation at all and 10 means extremely unpleasant sensation, and finally (5) pain sensitivity around the wound using a thin, short length of plastic.

The length of time needed to take part in this study will depend on how long the wound care procedure takes. The time could be approximately 45 minutes to 60 minutes (1 hour) per visit and 90 minutes (1½ hour) to 120 minutes (2 hours) in total for the study because 2 days are needed to complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (≥ 21 years) have to have an open wound with duration of no more than 10 days that requires wound care
* be able to self-report their pain
* had a pain intensity score > 3 during previous wound care procedure
* has intravenous access

Exclusion Criteria:

* Patients with an injury that impairs sensation in the wound area according to a medical diagnosis
* has an allergy to morphine or ketamine
* has not received morphine previously
* In addition, patients who are 65 years of age or older.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Puntillo, RN, DNSc, Study Chair — Regents of the University of California, San Francisco
Locations (2):
- University of California San Francisco, San Francisco, California, United States
- Trauma Hospital Puerto Rico Medical Center, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arroyo-Novoa CM, Figueroa-Ramos MI, Miaskowski C, Padilla G, Paul SM, Rodriguez-Ortiz P, Stotts NA, Puntillo KA. Efficacy of small doses of ketamine with morphine to decrease procedural pain responses during open wound care. Clin J Pain. 2011 Sep;27(7):561-6. doi: 10.1097/AJP.0b013e318211936a. PMID 21436683

RESULTS

PARTICIPANT FLOW:
Groups:
- Morphine Plus Ketamine, Then Morphine Plus Saline: During the first wound care procedure, patients received morphine 0.05 mg/kg (a maximum dose of 4 mg) plus ketamine 0.25 mg/kg. Then, during the second wound care procedure, they were cross-over to receive morphine 0.1 mg/kg plus Saline.
- Morphine Plus Saline, Then Morphine Plus Ketamine: During the first wound care procedure, patients received morphine 0.1 mg/kg (a maximum dose of 8 mg) plus saline. Then, they were cross-over to receive morphine 0.05 mg/kg (a maximum dose of 4 mg) plus ketamine 0.25 mg/kg.
Period: Overall Study
Arm/Group | Morphine Plus Ketamine, Then Morphine Plus Saline | Morphine Plus Saline, Then Morphine Plus Ketamine
Started | 7 | 5
Completed | 7 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Morphine Plus Ketamine First: During the first wound care procedure, patients received morphine 0.05 mg/kg (maximum dose of 4 mg) plus ketamine 0.25 mg/kg. Then, during the second wound care procedure, they received morphine 0.1 mg/kg (maximum dose of 8 mg) plus saline.
- Morphine Plus Saline First: During the first wound care procedure, patients received morphine 0.1 mg/kg (maximum dose of 8 mg) plus saline. Then, during the second wound care procedure, they received morphine 0.05 mg/kg (maximum dose of 4 mg) plus ketamine 0.25 mg/kg.
- Total: Total of all reporting groups
Arm/Group | Morphine Plus Ketamine First | Morphine Plus Saline First | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (9.6) | 32.5 (4.4) | 32.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: The degree of pain described by participants on a numeric rating scale of 0 to 10, where 0 = no pain and 10 = worst pain imaginable
Time Frame: Immediately after the wound care procedure
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Morphine Plus Ketamine: Participants who received morphine 0.05 mg/kg (a maximum dose of 4 mg) plus ketamine 0.25 mg/kg IV in either the first or second wound care procedure.
- Morphine Plus Saline: Participants who received morphine 0.1 mg/kg (a maximum dose of 8 mg) plus saline IV in either the first or second wound care procedure.
Arm/Group | Morphine Plus Ketamine | Morphine Plus Saline
Number analyzed (Participants) | 11 | 11
score on a scale | 3.1 (.99) | 6.8 (.92)

2. Secondary Outcome: Wound Pain Quality
Description: Short-form McGill Pain Questionnaire. The questionnaire has 15 adjectives to describe the pain. Each is rated on a 4-point scale (i.e., none, mild, moderate, or severe. Total wound pain quality score can range from 0 to 45.
Time Frame: Immediately after the procedure
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Morphine Plus Ketamine: Participants who received morphine 0.05 mg/kg (maximum dose of 4 mg) plus ketamine 0.25 mg/kg in either the first or second wound care procedure.
- Morphine Plus Saline: Participants who received morphine 0.1 mg/kg (maximum dose of 8 mg) plus saline in either the first or second wound care procedure.
Arm/Group | Morphine Plus Ketamine | Morphine Plus Saline
Number analyzed (Participants) | 11 | 11
units on a scale | 13.6 (3.6) | 17.6 (3.7)

ADVERSE EVENTS:
Groups:
- Morphine Plus Ketamine: Patients received morphine 0.05 mg/kg (maximum dose of 4 mg) plus ketamine 0.25 mg/kg (MK) during the first or second wound care procedure according to randomization
- Morphine Plus Saline: Patients received morphine 0.1 mg/kg (maximum dose of 8 mg) plus saline (MS) during the first or second wound care procedure according to randomization
Arm/Group | Morphine Plus Ketamine | Morphine Plus Saline
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 10/11 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine Plus Ketamine (N=11) | Morphine Plus Saline (N=11)
strange sensations (Nervous system disorders) | 10 (10) | 0 (0) — Patients reported strange, unpleasant sensations.

LIMITATIONS AND CAVEATS:
The sample size was small, and all patients were male. Blinding was challenging to assure when patients demonstrated adverse effects associated with ketamine. In addition, because different orthopedic technicians performed the WCPs, the effect of the variability in the procedure technique on pain could not be controlled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes